CLINICAL TRIAL: NCT02371954
Title: Exercise to Prevent Depression and Anxiety in Older Hispanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Daniel Enrique Jimenez, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20140607
Record Dates: First submitted 2015-01-21; First posted 2015-02-26 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Health Promotion (Experimental): Happy Older Latinos are Active (HOLA) is multicomponent health promotion intervention led by a community health worker (CHW). First component is a social and physical activation session. Participants meet individually with CHW for 30 minutes once at week 1, then again at week 8 (the midway point). Second component is a moderate intensity group walk. Groups will consist of 6 participants and will meet for one hour, 3 times a week, for 16 weeks. Third component is pleasant events scheduling during cool down phase of the group walk.
  Interventions: Behavioral: Happy Older Latinos are Active
- Psychoeducation (Active Comparator): Participants will be given a fotonovela and will meet once a month after they receive the fotonovela to discuss their thoughts on the materials they received. These discussion groups will last one hour and will consist of 10 participants.
  Interventions: Other: Fotonovela

INTERVENTIONS:
Behavioral: Happy Older Latinos are Active — Health promotion intervention desgined to prevent anxiety and depression in at risk older Hispanics
  Other Names: HOLA
  Arms: Health Promotion
Other: Fotonovela — Comic book style informational booklet designed for people with low literacy to educate them on mental illness.
  Arms: Psychoeducation

SUMMARY:
The study is a randomized pilot trial of a health promotion intervention in the prevention of anxiety and depression in older Hispanics.

DETAILED DESCRIPTION:
Eligible participants will be randomized to either the Happy Older Latinos are Active (HOLA) intervention or a psychoeducation condition. Participants randomized to HOLA will participate in a group exercise, 3 times a week, for 16 weeks. The exercise is a moderate intensity walk at a centrally located park in Miami-Dade county and will last for an hour (10 minute warmup/stretching, 30 minute walk, 5 minute cool down). Groups will consist of 6 participants and be led by a community health worker. During the cool down phase, participants will plan a pleasant event to be done in between sessions. Participants randomized to the psychoeducation component will receive a fotonovela and will meet once a month after they receive the fotonovela to discuss their thoughts on the materials they received. These discussion groups will last one hour and will consist of 10 participants. A total of 60 participants will be randomized (30 to HOLA, 30 to fotonovela). Assessments will be conducted at baseline, post intervention, 6 months post-intervention, and 12 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Hispanic (self-identified);
2. Age 60+;
3. Minor depression as defined by a primary DSM-IV Axis I diagnosis of minor depressive disorder or subthreshold depression defined as a score ≥ 3 on the Patient Health Questionnaire (PHQ-2), OR subthreshold anxiety as defined as a score ≥ 3 on the Generalized Anxiety Disorder-2 scale (GAD-2);
4. Absence of episodes of major depression and anxiety disorders for past 12 months (as determined by the MINI);
5. Voluntary informed consent for participation in the study by the participant or by the participant's legally designated guardian or conservator;
6. Medical clearance for participation in an exercise program by a physician, physician's assistant, or nurse practitioner;
7. Expect to be resident in Miami for the subsequent 12 months.

Exclusion Criteria:

1. Currently residing in a nursing or group home;
2. A terminal physical illness expected to result in the death within one year;
3. A diagnosis of dementia, co-morbid diagnosis of dementia, or significant cognitive impairment as indicated by an MMSE score <24;
4. Presence of any axis 1 psychiatric disorder or substance abuse during preceding 12 months;
5. History of psychiatric disorders other than non-psychotic unipolar major depression or anxiety disorder;
6. High suicide risk, i.e., intent or plan to attempt suicide in the near future (a response of "yes" to questions 3, 4, and/or 5 on the Paykel Questionnaire);
7. Participants taking cognitive enhancing medication or psychotropic medications (e.g. antidepressants);
8. unable to complete 400 m walk test in less than 15 min;
9. if participant heart rate exceeded 170 beats per minute OR systolic blood pressure exceeds 180 during 400 m walk test;
10. chest or leg pain, dyspnea, dizziness, feeling faint, or other significant symptoms while completing 400 m walk test;

(i) acute or severe medical illness that would prevent participants from walking at a moderate pace for 45 minutes, three times a week.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Prevention of major depression, generalized anxiety, and social anxiety as measured the Mini International Neuropsychiatric Interview | change from baseline at 16 months
  I will be using the Mini International Neuropsychiatric Interview to test whether the HOLA intervention was successful in preventing participants from getting major depressive disorder, generalized anxiety disorder, and social anxiety disorder.

SECONDARY OUTCOMES:
Physical functioning as measured by the World Health Organization Disability Assessment Schedule 2.0 (WHO-DAS 2) | change from baseline at 16 months
  I will be measuring the effect the HOLA intervention has on the scores of the Getting Around, Life Activities, and Self-Care subscales of the WHO-DAS 2.0
Social functioningas measured by the World Health Organization Disability Assessment Schedule 2.0 (WHO-DAS 2) | change from baseline at 16 months
  I will be measuring the effect the HOLA intervention has on the scores of the Getting Along with People and Participation in Life subscales of the WHO-DAS 2.0
Self-efficacy as measured by the General Self-Efficacy Scale | change from baseline at 16 months
  I will be measuring the effect the HOLA intervention has on total scores of the General-Self Efficacy Scale.
Sleep quality as measured by the Pittsburgh Sleep Quality Index | change from baseline at 16 months
  I will be measuring the effect the HOLA intervention has on the total scores of the Pittsburgh Sleep Quality Index
Change in depression symptom severity as measured by the Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR). | change from baseline at 16 months
  I will be measuring the effect the HOLA intervention has on the total scores of the QIDS-SR
Change in anxiety symptom severity as measured by the Beck Anxiety Inventory (BAI) | change from baseline at 16 months
  I will be measuring the effect the HOLA intervention has on the total scores of the BAI

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Jimenez, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Mental Health Hospital, Miami, Florida, United States

REFERENCES:
- [Derived] Jimenez DE, Ross EJ, Weinstein ER, Martinez Garza D, Signorile JF, Perdomo-Johnson D, Martinez C. "Caminando y socializando con Happy Older Latinos are Active (HOLA)": Results of a randomized clinical trial to promote health and prevent depression and anxiety in older Latinos. J Consult Clin Psychol. 2025 Apr;93(4):317-327. doi: 10.1037/ccp0000923. Epub 2024 Dec 2. PMID 39621372
- [Derived] Jimenez DE, Reynolds CF 3rd, Alegria M, Harvey P, Bartels SJ. The Happy Older Latinos are Active (HOLA) health promotion and prevention study: study protocol for a pilot randomized controlled trial. Trials. 2015 Dec 18;16:579. doi: 10.1186/s13063-015-1113-3. PMID 26683695